CLINICAL TRIAL: NCT02095249
Title: Hypoxia and Stem Cell Content as Aggression Factors in Prostate Cancer
Brief Title: Prostate Hypoxia - TIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UHN REB 13-7172-C
Record Dates: First submitted 2014-03-12; First posted 2014-03-24 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pimonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pimonidazole (Other)
  Interventions: Drug: Pimonidazole

INTERVENTIONS:
Drug: Pimonidazole — Pimonidazole is to be administered to patients scheduled for radical prostatectomy one day prior to surgery.

SUMMARY:
Prostate cancer is the most commonly diagnosed form of cancer in Canadian men. In 2006, greater than 250,000 men were diagnosed with prostate cancer in the United States and Canada with more than 32,000 men dying of their disease. Using the prognostic variables of T-category, the serum prostate specific antigen (PSA), and the pathologic Gleason score (GS), men with localized prostate cancer are placed in low, intermediate and high-risk groupings. Usually this is treated with surgery, radiation therapy, hormone therapy and/or watchful waiting (also known as active surveillance). While these treatments are quite effective, tumours are likely to recur in about 40% of cases. There is a need for additional prostate cancer treatments. To address this need, many experimental therapies are being developed and tested in mice with prostate tumors. This includes the study of aggressive prostate cancer cells such as stem cells, or Tumour Initiating Cells (TICs), or oxygen deprived cells, which may be the ones most likely to re-grow into a tumour or spread throughout the body. Researchers want to try and isolate these special cells from the prostate after surgery to study their features, and to see if they can re-grow as solid tumours in mice. Researchers would like to test whether the prostate cancer stem cells are more resistant or less resistant to treatments. This will allow researchers to study and test new treatments that specifically target resistant and aggressive prostate cancer cells. The investigators hypothesize that marker-defined TIC cells or hypoxic cancer cells have unique genetics in primary prostate cancers and are relatively chemo- and radio-resistant.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients with bulky intermediate risk or high-risk disease who have already agreed to undergo an open radical prostatectomy at Princess Margaret Cancer Centre-UHN:
* Clinical stage T2-T3 N0 M0
* Pathology of adenocarcinoma of the prostate AND
* Gleason score 7 with >/= 50 % biopsies involved with tumour; OR
* Gleason score 8 or above (any percentage of biopsies)

Exclusion Criteria:

* Patients with clinical T4, N1 or M1 disease
* Patients with histologies other than adenocarcinoma
* Patients unable to ingest pimonidazole tablets

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Quantitation of pimonidazole staining (a.u./cm2) in radical prostatectomy specimens as determinant of biochemical failure | 3 years
  Radical prostatectomy specimens will stained for pimonidazole uptake using antibody-based immunofluorescence assays

SECONDARY OUTCOMES:
Quantitation of tumour initial cells by immunohistochemistry (cells/mm2) in radical prostatectomy specimens as determinant of biochemical failure | 3 years
  Radical prostatectomy specimens will stained for cell surface markers pertaining to tumor initiating cells using immunofluorescence assays

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Berlin, MD., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada